CLINICAL TRIAL: NCT06879886
Title: MRD-Guided Surveillance in Resectable Stage IV Metastatic Colorectal Cancer (SURVEILLANCE-II)
Acronym: SURII
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery Department, Zhongshan hospital, Fudan University, Fudan University
Other Study IDs: SURVEILLANCE-II
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC); Colorectal Cancer Liver Metastases (CRLM)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — In this study, the specific types of samples that will be retained are peripheral blood samples collected from patients at multiple time points. These samples will be used for circulating tumor DNA (ctDNA) analysis to assess minimal residual disease (MRD) status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MRD-Guided Surveillance in Resectable Stage IV Metastatic Colorectal Cancer

SUMMARY:
This study aims to explore the relationship between minimal residual disease (MRD) status and disease recurrence in patients with resectable stage IV metastatic colorectal cancer (mCRC). MRD refers to the presence of cancer cells that remain in the body after treatment but are undetectable by traditional imaging methods. The study will use a blood-based circulating tumor DNA (ctDNA) methylation test to assess its ability to predict cancer recurrence and survival outcomes.

Patients who are newly diagnosed with resectable stage IV mCRC and have not yet received any treatment will be enrolled. Blood samples will be collected at multiple time points, including before surgery, after surgery, and during follow-up visits over two years. The study will compare MRD status with recurrence-free survival (RFS), overall survival (OS), and the time it takes for MRD to detect recurrence compared to standard imaging methods.

The goal is to determine whether MRD monitoring can provide an early warning of cancer recurrence and help guide treatment decisions. This study may offer valuable insights into improving postoperative surveillance and personalized treatment strategies for metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study designed to evaluate the effectiveness of ctDNA-based MRD monitoring in predicting disease recurrence and survival outcomes in patients with resectable stage IV metastatic colorectal cancer (mCRC). The study will enroll 181 patients who have not previously received chemotherapy, radiotherapy, or targeted therapy.

Key Objectives

Primary Objective:

To explore the correlation between MRD status and recurrence-free survival (RFS) in resectable stage IV mCRC patients.

Secondary Objectives:

To assess the relationship between MRD status and 1-year/2-year event-free survival (1yEFS, 2yEFS).

To evaluate the association between MRD status and 2-year recurrence-free survival (2yRFS).

To assess the impact of MRD status on overall survival (OS).

Exploratory Objective:

To determine the average time by which MRD detection precedes imaging-based detection of disease recurrence.

Study Design

Patients will undergo blood sampling at key time points:

Baseline (pre-treatment) Pre-surgery (0-7 days before surgery) Post-surgery (7±2 days after surgery) Follow-up visits at 1, 3, 6, 9, 12, 18, and 24 months post-surgery MRD status will be assessed using a ctDNA methylation-based PCR test, which provides a rapid, cost-effective alternative to traditional NGS-based methods.

Statistical Analysis Kaplan-Meier survival analysis will be used to estimate RFS, EFS, and OS. Cox proportional hazards models will assess whether MRD status serves as an independent prognostic factor for recurrence.

Multivariate analysis will adjust for clinical variables, including tumor burden and treatment history.

Ethical Considerations The study adheres to the principles of the Declaration of Helsinki and Chinese Good Clinical Practice (GCP) guidelines.

Informed consent will be obtained from all participants, and privacy and confidentiality will be strictly maintained.

Expected Outcomes This study aims to validate the clinical utility of ctDNA-based MRD monitoring in predicting recurrence and survival outcomes for resectable stage IV mCRC patients. If successful, MRD testing may offer a more effective tool for postoperative surveillance and treatment planning, allowing for earlier interventions and improved long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, male or female;
2. histologically confirmed primary foci of colorectal adenocarcinoma (i.e., adenoepithelial carcinoma, including adenocarcinoma, mucinous adenocarcinoma, imprinted cell carcinoma, and undifferentiated carcinoma; excluding adenosquamous carcinoma); (3) Preoperative stage IV and no surgical resection; (4) Not receiving chemotherapy, radiotherapy, targeted therapy or other anti-tumor therapy;

5) Surgical resection of primary/metastatic foci is possible; 6) ECOG score 0-1; 7) Subjects voluntarily enrolled in the study and signed the informed consent, good compliance, and actively cooperate with the regular clinical follow-up clinic back in the hospital.

Exclusion Criteria:

1. Previous other malignant tumors (including non-adenocarcinoma colorectal cancer);
2. Pregnant and lactating women;
3. Patients with other concurrent illnesses that, in the judgment of the investigator, may interfere with follow-up and short-term survival;
4. The subject has other factors that may cause this study to be forced to be terminated halfway, such as other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors that would affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with resectable stage IV metastatic colorectal cancer (mCRC) who have not received prior systemic treatment. Participants will be recruited from multiple clinical centers and must meet specific eligibility criteria to ensure the study's validity.
  Key Characteristics of the Study Population:
  Diagnosis: Histologically confirmed colorectal adenocarcinoma (including adenocarcinoma, mucinous adenocarcinoma, signet-ring cell carcinoma, and undifferentiated carcinoma; excluding adenosquamous carcinoma).
  Stage: Clinical stage IV disease, confirmed by preoperative imaging and clinical assessment as having resectable primary and metastatic lesions.
  Treatment History: No prior chemotherapy, radiotherapy, targeted therapy, or other anti-cancer treatments.
  Surgical Eligibility: Candidates must be eligible for curative-intent resection of both the primary tumor and metastatic lesions.
  General Health Status: ECOG performance status 0-1, indicating
Sampling Method: Non-Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Exploring the correlation between MRD status and rate of disease recurrence (RFS) in people with stage IV metastatic resectable colorectal cancer | From surgery to disease recurrence or up to 24 months
  Exploring the correlation between MRD status and rate of disease recurrence (RFS) in people with stage IV metastatic resectable colorectal cancer

SECONDARY OUTCOMES:
Correlation of MRD status with 1-year event-free survival (1yEFS) | From surgery to 12 months
  Correlation of MRD status with 1-year event-free survival (1yEFS)
Correlation of MRD status with 2-year event-free survival (2yEFS) | From surgery to 24 months
  Correlation of MRD status with 2-year event-free survival (2yEFS)
Correlation of MRD status with 2-year recurrence-free survival (2yRFS) | From surgery to 24 months
  Correlation of MRD status with 2-year recurrence-free survival (2yRFS)
Correlation of MRD status with overall survival (OS) | From surgery to death or up to 24 months
  Correlation of MRD status with overall survival (OS)

OTHER OUTCOMES:
MRD detects disease recurrence earlier than imaging (CT) average advance time | From surgery to disease recurrence, assessed up to 24 months
  MRD detects disease recurrence earlier than imaging (CT) average advance time

IPD SHARING:
Plan to Share IPD: No